CLINICAL TRIAL: NCT05029310
Title: Effects of Patiromer on Pharmacokinetics of Immunosuppresive Drugs in Renal Transplant Recipients
Acronym: TACPAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Geir Mjøen, Resident, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 148684
Record Dates: First submitted 2021-08-26; First posted 2021-08-31 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Hyperkalemia; Kidney Transplant
Keywords: kidney transplant; Hyperkalemia
MeSH Terms: conditions — Hyperkalemia

STUDY DESIGN:
Intervention Model Description: Patients already taking tacrolimus start treatment with patiromer. After seven days tacrolimus kinetics are studied. Seven days after discontinuation of patiromer, tacrolimus kinetics are repeated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All patients use both patiromer and tacrolimus (Experimental): Pharmacokinetic investigation of tacrolimus performed in both the presence and absence of patiromer for all patients.
  Interventions: Drug: Patiromer Oral Product

INTERVENTIONS:
Drug: Patiromer Oral Product — interaction study

SUMMARY:
Patiromer lowers potassium effectively in patients with hyperkalemia and chronic kidney disease. Patients with a kidney transplant usually have reduced renal function and may also develop hyperkalemia. However, potential interactions between immunosuppressive medications and patiromer have not been evaluated. These interactions could involve change in AUC of immunosuppressive drugs, such as calcineurin inhibitors or mycophenolate, or increased risk of hypomagnesemia, since both tacrolimus and patiromer have this potential side effect. We wish to evaluate potential interactions to ensure safe use of this drug in the transplant population.

DETAILED DESCRIPTION:
Patients with a kidney transplant may develop hyperkalemia. This could be due to different mechanisms. In some patients it could be due to reduced kidney function. In others, it could be secondary to renal tubular acidosis type 4 caused by necessary medications used after transplantation.

The most important medicines contributing to hyperkalemia after kidney transplantation are calcineurin inhibitors which are a compulsory part of the immunosuppressive regimen, ACE inhibitors or ARBs in patients with hypertension, and trimethoprim-sulfa, which is used as infection prophylaxis in all patients during the first 6 months after transplantation. In the weeks after renal transplantation around 5-10% of transplant patients at our institution at some point develop hyperkalemia above the limit where some type of management of hyperkalemia would be indicated. As the drugs mentioned above can rarely or not at all be withdrawn after transplantation, most doctors will either observe the hyperkalemia untreated or try to lower the potassium level.

In outpatients with s-potassium of 5 - 6.5, urgent management is usually not necessary. However, some kind of intervention is still indicated, to make sure that the potassium will decrease during the next days. Patiromer could be an interesting alternative in those kidney transplanted patients that are in this category. We are not aware of any published studies describing the use of patiromer in the transplant population. We intend to investigate if there is any pharmacokinetic interaction between patiromer and immunosuppressive drugs affecting the blood concentration of the latter.

ELIGIBILITY:
Inclusion Criteria:

1. Renal transplant recipients, at least 3 weeks after transplantation, who receive Tacrolimus as part of their immunosuppressive therapy, with stabile tacrolimus dose and trough tacrolimus concentration.
2. Recipients 18 years of age or older.
3. Hyperkalemia (K>5 and <6,0)
4. Signed informed consent.

Exclusion Criteria:

1. Concomitant treatment with: diltiazem, verapamil, fenytoin, carbamazapin, fluconazole, ketoconazole, vorikonazole, erythromycin, clarithromycin, resonium-calcium, and/or sodium zirconium cyclosilicate.
2. Constipation, defined as fewer than three bowel movements per week.
3. Hypomagnesemia less than 0.6 mmol/L.
4. Serum potassium level of greater than 6.0 mEq/L.
5. Increased immunologic risk patient (DSA, ABO-incompatible transplant).
6. Pregnancy or suspected pregnancy (pregnancy is excluded at time of transplantation by measuring HCG, kidney transplanted patients should not become pregnant before at least one year after transplant, and no transplanted patient has ever become pregnant during the first weeks after transplantation. They are all informed regarding different types of contraception). Fertile women will be tested for pregnancy before inclusion.
7. Hypersensitivity/allergy to patiromer.
8. Other serious medical or psychiatric condition likely to interfere with participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
study potential interaction between patiromer and tacrolimus | two weeks
  Log-transformed AUC0-tau of tacrolimus between patiromer vs. no patiromer

SECONDARY OUTCOMES:
Determine effect of patiromer on potassium concentration. | two weeks
  Delta-value change of serum potassium from start of treatment to 7 days after start of treatment, and delta-value change of serum potassium from 7 days after start of treatment to 7 days after end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Geir Mjøen, MD, Principal Investigator — MD
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
no plan